CLINICAL TRIAL: NCT02619292
Title: Mindful Movement for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint John's Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMP-001
Record Dates: First submitted 2015-11-06; First posted 2015-12-02 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: cancer survivor; immune function
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindful Movement Program (Experimental): Mindfulness is "moment-to-moment, present-centered, purposive non-judgmental awareness"; Dance/movement therapy is a multidimensional approach that integrates body awareness, expression and acceptance to facilitate physical, emotional, cognitive, social and spiritual integration of individuals
  Interventions: Behavioral: Mindful Movement Program

INTERVENTIONS:
Behavioral: Mindful Movement Program — Mindfulness is turning one's awareness to the present moment. Movement-dance therapy is the expression of thoughts or feelings through body movement, under the supervision of a licensed professional.

SUMMARY:
The purpose of this study is to determine if participating in a Mindful Movement Program (MMP) (learning how to be mindful in one's movement), positively affects the body's immune functions improves mindfulness and reduces worries about cancer returning. All participants will be in this study about three months.

DETAILED DESCRIPTION:
Breast cancer survivors (BCS) may experience psychological and physical effects long after treatment is over. Some research shows that practicing mindfulness, and movement types of activities such as qi gong or yoga may lead to improvements in emotional and physical well-being, including improved immune function. Immune function can be negatively affected by stress and worry, and this has an unknown effect on the risk of cancer recurrence. Psychological and physical interventions that help enhance an individual's wellbeing and reduce stress and worry may have a positive influence on immune function and in turn, reduce the risk of cancer recurrence. While there is limited research in this area, and none with dance therapy, little attention has been given to older BCS. However, understanding of immune function suggests that older women may be the best group to target for such interventions. Previous research with BCS age 50 or older who participated in a 12-week program combining mindfulness practice with dance/movement therapy (Mindful Movement Program) demonstrated positive effects: participants were more mindful in their day-to-day living and had less worry about the cancer coming back. Participants also reported through focus groups that the Mindful Movement Program (MMP) had improved their overall well-being. No laboratory tests of the body's immune response to MMP were included.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed at age 50 or older with stage 0-III disease
* 6 months or more since completion of primary breast cancer treatment
* have a medical release from their physician
* English-speaking
* not pregnant
* no weekly practice of yoga, qi gong, tai chi, dance/movement therapy, or mindfulness meditation practice

Exclusion Criteria:

* Males with breast cancer

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Immune markers | 18 weeks
  Improvement in serum markers of immune cell phenotype at week 18

SECONDARY OUTCOMES:
Mindful Movement Intervention Experience | 18 weeks
  Improvement in mindfulness attitude as measured on Meditative Movement Inventory (MMI)
Mindful Movement Intervention Experience | 18 weeks
  Improvement in mindfulness attitude as measured on Perceived Exertion Scale (PES)
Mindful Movement Intervention Experience - Mindfulness Intention | 18 weeks
  Improvement in mindfulness attitude as measured on Mindfulness Intention (modified from Segal, 1-item)

OTHER OUTCOMES:
Fear of Recurrence | 18 weeks
  Fear of recurrence as measured on Fear of Recurrence (FOR) scale
Mindfulness attention | 18 weeks
  Improvement in mindfulness attitude as measured with the Mindful Attention Awareness Scale (MAAS)
Mindfulness attitude | 18 weeks
  Improvement in mindfulness attitude as measured with the Experiences Questionnaire (EQ)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Crane-Okada, PhD, RN, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- Margie Petersen Breast Center at Providence Saint John's Health Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided